CLINICAL TRIAL: NCT03167528
Title: Contribution of Learning and Practice of Different Complementary Therapies in Pulmonary Transplant Patients
Acronym: TOOLBOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016/59; 2016-A01654-47 (Other: ANSM)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Lung Transplant
Keywords: Pain; Quality of life
MeSH Terms: conditions — Pain | interventions — Hypnosis; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung transplant (Experimental): Patients who must undergo a lung transplant at the FOCH hospital.
  Before and after transplantation, patients benefits of learning and realization sessions of complementary techniques:
  * Relaxation,
  * Hypnosis,
  * Holistic gymnastics,
  * Transcutaneous electrical nerve stimulation (TENS),
  * Sophrology.
  Interventions: Behavioral: Relaxation; Behavioral: Hypnosis; Behavioral: Holistic gymnastics; Device: Transcutaneous electrical nerve stimulation (TENS); Behavioral: Sophrology

INTERVENTIONS:
Behavioral: Relaxation — Relaxation
Behavioral: Hypnosis — Hypnosis
Behavioral: Holistic gymnastics — holistic gymnastics
Device: Transcutaneous electrical nerve stimulation (TENS) — TENS
Behavioral: Sophrology — Sophrology

SUMMARY:
The aim of the study is to evaluate, 3 months after lung transplantation, integration and appropriation by the patient of complementary techniques (" Toolbox " included relaxation, autohypnosis, relaxation therapy, TENS (if pain) and holistic gymnastics to improve the comfort and the quality of life in very high-technology care pathway

DETAILED DESCRIPTION:
Patients approaching a lung transplant will face specific infectious, immunological, ventilatory and hemodynamic problems but also to painful, stressful and anxiety-provoking situations. Learning different complementary therapies in the pre-transplant period allows patients to have personal tools to improve their comfort before and after the transplant. These tools can be used by patients who have acute or chronic pain symptoms, to support painful examination or care, and for situations of stress and anxiety.

The project aims to present different therapies complementary to patients. Before and after transplant, patients benefits of learning and realization sessions of these techniques. They appropriate the techniques and choose the ones that suit best.

The overall benefit will be judged comparing period before transplant to period after transplant on different criteria.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for a lung transplantation benefiting from a pre-transplant evaluation

Exclusion Criteria:

* transplant patient in emergency
* delay between pre-transplant evaluation and transplantation over 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Number of sessions of complementary techniques | 3 months
  Number of sessions of complementary techniques practiced by the patient alone and by the patient with an investigator of the team.

SECONDARY OUTCOMES:
Implication and satisfaction degree measured by Visual Analogical Scale (VAS) | 3 months
  Implication and satisfaction of the patient regarding the different techniques. Investment, autonomy, conformity to instructions, adaptation to different situation and use of the different techniques are evaluated by the patient and by the investigators using 5 Visual Analogical Scales (VAS)
Efficacy of complementary techniques on the pain felt. | 3 months
  Evaluate the efficacy of the "toolbox" on presence, intensity, location, type of pain 3 months after transplant by VAS, questionnaire DN4 and Kehlet's questionnaire.
  3 VAS to measures the intensity of pain on a scale of 0 (no pain) to 10 (worst possible pain), and 1 question to locate the pain.
  DN4 to identify neuropatic pain: 4 questions to answer by "yes" or "no". "yes" = 1 point, "no" = 0 point. Total score ≥ 4/10 = positive test.
  Kehlet's questionnaire to evaluate the impact of pain on activities.
Efficacy of complementary techniques on anxiety and depression level | 3 months
  Evaluate the efficacy of the "toolbox" on anxiety and depression level 3 months after transplant by Hospital Anxiety and Depression (HAD) scale. 14 items rated from 0 to 3. Seven questions relate to anxiety and seven others to the depression. Two scores (maximum of each score = 21).
Efficacy of complementary techniques on stress level | 3 months
  Evaluate the efficacy of the "toolbox" on stress level 3 months after transplant by Perceived Stress Scale. 10 items rated from 0 to 5.
  Total score < 21 = someone who knows how to manage stress. Total score between 21 and 26 = someone who usually knows how to manage stress, except in certain situations.
  Total score > 27 = someone who don't knows how to manage stress.
Efficacy of complementary techniques on sleep quality | 3 months
  Evaluate the efficacy of the "toolbox" on sleep quality 3 months after transplant by Spiegel sleep score. 6 items rated from 0 to 5.
  More the score is lower, more the sleep disorders is serious.
Efficacy of complementary techniques on quality of life | 3 months
  Evaluate the efficacy of the "toolbox" on quality of life 3 months after transplant by questionnaire Quality of life EuroQol - 5 Dimension (EQ5D) and the EuroQol Visual Analogue scale (EQ VAS) .
  EQ5D: 5 dimensions. Each dimension has 3 levels: no problems, some problems, extreme problems.
  EQ VAS: records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille MICHEL-CHERQUI, MD, Principal Investigator — FOCH Hospital
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ringsted TK, Wildgaard K, Kreiner S, Kehlet H. Pain-related impairment of daily activities after thoracic surgery: a questionnaire validation. Clin J Pain. 2013 Sep;29(9):791-9. doi: 10.1097/AJP.0b013e318278d4e2. PMID 23370071
- [Background] Bouhassira D, Lanteri-Minet M, Attal N, Laurent B, Touboul C. Prevalence of chronic pain with neuropathic characteristics in the general population. Pain. 2008 Jun;136(3):380-387. doi: 10.1016/j.pain.2007.08.013. Epub 2007 Sep 20. PMID 17888574
- [Background] Lepine JP, Godchau M, Brun P, Lemperiere T. [Evaluation of anxiety and depression among patients hospitalized on an internal medicine service]. Ann Med Psychol (Paris). 1985 Feb;143(2):175-89. No abstract available. French. PMID 4037594
- [Background] Lesage FX, Berjot S, Deschamps F. Psychometric properties of the French versions of the Perceived Stress Scale. Int J Occup Med Environ Health. 2012 Jun;25(2):178-84. doi: 10.2478/S13382-012-0024-8. Epub 2012 Apr 19. PMID 22528542
- [Background] Spiegel R. Sleep and sleeplessness in advanced age. Advances in Sleep Research. Lancaster UK: MTP Press; 1981. p. 1-272.
- [Background] Michel-Cherqui M, Ley L, Szekely B, Dreyfus JF, Fischler M. Prevalence and characteristics of pain in patients awaiting lung transplantation. J Pain Symptom Manage. 2015 Mar;49(3):548-54. doi: 10.1016/j.jpainsymman.2014.07.011. Epub 2014 Aug 21. PMID 25150816
- [Background] Wildgaard K, Iversen M, Kehlet H. Chronic pain after lung transplantation: a nationwide study. Clin J Pain. 2010 Mar-Apr;26(3):217-22. doi: 10.1097/AJP.0b013e3181b705e4. PMID 20173435
- [Background] Girard F, Chouinard P, Boudreault D, Poirier C, Richard C, Ruel M, Ferraro P. Prevalence and impact of pain on the quality of life of lung transplant recipients: a prospective observational study. Chest. 2006 Nov;130(5):1535-40. doi: 10.1378/chest.130.5.1535. PMID 17099034
- [Background] Gross CR, Kreitzer MJ, Thomas W, Reilly-Spong M, Cramer-Bornemann M, Nyman JA, Frazier P, Ibrahim HN. Mindfulness-based stress reduction for solid organ transplant recipients: a randomized controlled trial. Altern Ther Health Med. 2010 Sep-Oct;16(5):30-8. PMID 20882729
- [Background] Goldbeck L, Fidika A, Herle M, Quittner AL. Psychological interventions for individuals with cystic fibrosis and their families. Cochrane Database Syst Rev. 2014 Jun 18;2014(6):CD003148. doi: 10.1002/14651858.CD003148.pub3. PMID 24941199
- [Background] 13. Servant D. La relaxation, nouvelles approches nouvelles pratiques: Elsevier-Masson; 2009.
- [Background] McCraty R, Zayas MA. Cardiac coherence, self-regulation, autonomic stability, and psychosocial well-being. Front Psychol. 2014 Sep 29;5:1090. doi: 10.3389/fpsyg.2014.01090. eCollection 2014. PMID 25324802
- [Background] Sarabia-Cobo CM. Heart coherence: a new tool in the management of stress on professionals and family caregivers of patients with dementia. Appl Psychophysiol Biofeedback. 2015 Jun;40(2):75-83. doi: 10.1007/s10484-015-9276-y. PMID 25796509
- [Background] Anbar RD. Self-hypnosis for patients with cystic fibrosis. Pediatr Pulmonol. 2000 Dec;30(6):461-5. doi: 10.1002/1099-0496(200012)30:63.0.co;2-4. PMID 11109057
- [Background] Jensen MP. Hypnosis for chronic pain management: a new hope. Pain. 2009 Dec;146(3):235-237. doi: 10.1016/j.pain.2009.06.027. Epub 2009 Jul 10. No abstract available. PMID 19596518
- [Background] Tefikow S, Barth J, Maichrowitz S, Beelmann A, Strauss B, Rosendahl J. Efficacy of hypnosis in adults undergoing surgery or medical procedures: a meta-analysis of randomized controlled trials. Clin Psychol Rev. 2013 Jul;33(5):623-36. doi: 10.1016/j.cpr.2013.03.005. Epub 2013 Mar 26. PMID 23628907
- [Background] Carroll D, Moore RA, McQuay HJ, Fairman F, Tramer M, Leijon G. Transcutaneous electrical nerve stimulation (TENS) for chronic pain. Cochrane Database Syst Rev. 2001;(3):CD003222. doi: 10.1002/14651858.CD003222. PMID 11687055
- [Background] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Background] 21. Michel-Cherqui M. Effect of TENS (TransCutaneous Electrical NeuroStimulation) on post lung transplantation pain. 11th International Congress on Lung Transplantation Paris; 2014.